CLINICAL TRIAL: NCT06748872
Title: EPITOME-1015-I: a Phase I Study to Investigate the Safety, Tolerability and Preliminary Efficacy of a Third Generation TCR-T Therapy, MDG1015, in Epithelial Ovarian Carcinoma, Gastroesophageal (Junction) Adenocarcinoma, Myxoid (Round Cell) Liposarcoma And/or Synovial Sarcoma Subjects with Advanced Disease Expressing NY-ESO-1 And/or LAGE-1a
Brief Title: EPITOME-1015-I: a Study to Investigate the Safety and Tolerability of MDG1015 in Patients with Epithelial Ovarian Cancer, Gastroesophageal Adenocarcinoma, Round Cell Liposarcoma And/or Synovial Sarcoma
Acronym: EPITOME-1015-I
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medigene AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-TCR-004; 2024-516787-28-00 (EU CTIS Number); 2024-516787-28 (EudraCT Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Epithelial Ovarian Cancer; Gastro-esophageal Junction Cancer; Soft Tissue Sarcoma (STS); Myxoid Liposarcoma; Synovial Sarcoma
Keywords: TCR-T Therapy; dose escalation; Third Generation TCR-T Therapy; autologous, patient derived CD8+ T cells; single arm; open label; phase I; BOIN design; NY-ESO-1; LAGE-1a; solid tumors; PD1-41BB; Costimulatory Switch Protein; Armoring; Enhancement; First-in-human
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Sarcoma; Liposarcoma, Myxoid; Sarcoma, Synovial

STUDY DESIGN:
Intervention Model Description: Single arm, open label, multicenter, phase I study following a Bayesian optimal interval (BOIN) design for dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of MDG1015 (Experimental): MDG1015 is a first-in-class, 3rd generation TCR-T therapy consisting of autologous, patient-derived CD8+ T cells that are transduced with a New York esophageal squamous cell carcinoma-1 (NY-ESO-1)/ L antigen family member-1a (LAGE-1a)-specific, human leukocyte antigen (HLA)-A*02:01-restricted T cell receptor (TCR) and the costimulatory switch protein (CSP) programmed cell death protein 1 (PD1)-41BB administered following lymphodepletion chemotherapy.
  Interventions: Drug: Lymphodepletion; Biological: TCR-T cells (MDG1015)

INTERVENTIONS:
Drug: Lymphodepletion — Cylcophosamide and Fludarabine
Biological: TCR-T cells (MDG1015) — TCR-T cells (MDG1015)

SUMMARY:
MDG1015 is a third generation TCR-T therapy product targeting NY-ESO-1/LAGE-1a armored and enhanced by the PD1-41BB costimulatory switch protein (CSP). The study purpose is to establish the safety, tolerability and preliminary efficacy of MDG1015 in patients with epithelial ovarian cancer, gastroesophageal adenocarcinoma, round cell liposarcoma and/or synovial sarcoma that expresses NY-ESO-1 and/or LAGE-1a.

The main questions this clinical trial aims to answer are:

Can this TCR-T therapy MDG1015 be given to patients safely? What is the optimal dose of the TCR-T therapy MDG1015? If and what side effects do participants experience after receiving the TCR-T therapy MDG1015? Do participants experience a potential disease response after receiving the TCR-T therapy MDG1015?

Participants will:

Receive (in most cases) 1 single infusion of MDG1015 at a pre-defined dose level and will be followed up regularly up to 1 year. After one year, participants will enter the long term follow-up part up to 15 years after being treated. Any side effects and/or potential disease response will be documented during this period.

DETAILED DESCRIPTION:
The clinical study consists of screening, leukapheresis of mononuclear cells, LDC, followed by a single MDG1015 infusion on Day 0 and a subsequent hospitalization period of at least 3 days for in-patient safety monitoring. All Subjects who have received an MDG1015 infusion will continue to be followed regularly for safety and efficacy assessments in a post-treatment follow-up through month 12 (Y1) and long-term follow-up (LTFU) through years 2 - 15 in an out-patient setting. Dose Escalation Segment (DE) will evaluate an anticipated number of 4 dose levels to establish the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D). During the cohort expansion (CE) segment the MTD/RP2D will be confirmed

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ≥ 18 years of age and weigh ≥ 40 kg for Dose levels 1-3 and ≥ 50 kg for Dose level 4
2. Subject must have a confirmed diagnosis of either High grade serous or endometrioid ovarian, primary peritoneal or fallopian tube cancer Gastric or esophageal (junction) adenocarcinoma Myxoid (round cell) liposarcoma Synovial sarcoma
3. Subject's must have tested positive for HLA-A*02:01 genotype by a Sponsor designated central laboratory
4. Subject's tumor must have tested positive for NY-ESO-1 and/or LAGE-1a mRNA expression by a Sponsor designated central laboratory Both ≤1 year old archival tissue or fresh biopsy are allowed
5. Subjects diagnosed with an eligible indication must have exhausted treatment options with proven survival benefit
6. Subjects must have

   1. measurable disease
   2. Life expectancy ≥ 3 months per Investigator's opinion

8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 9. Adequate vital organ function 10. Adequate bone marrow function 11. Adequate coagulation profile 12. Toxicities from prior/ongoing therapies must have recovered to ≤ Grade 2 according to the CTCAE v5.0 or Subject's baseline excluding alopecia 14. Prior toxicities related to surgical procedures should have recovered to Grade ≤ 1 15. Women of childbearing potential (WCBP) or men who can father children must be willing and able to use adequate (e.g. barrier or licensed hormonal methods)

Exclusion Criteria:

1. Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined
2. HLA-A*02:02 or HLA-A*02:03 genotype
3. Pregnant or lactating women
4. Viral serology:

   1. Known infection with HIV-1/2, CMV (CMV required only for U.S. sites) or HTLV-1/2,
   2. Active infection with HBV or HCV
   3. Positive test for Mycoplasma or Treponema Pallidum
5. Uncontrolled infection(s) requiring intravenous anti-bacterial, anti-viral or anti-fungal treatment within 14 days prior to the first dose of LDC (patients receiving prophylactic antibiotics are eligible)
6. Inadequate venous access for or contraindications to leukapheresis
7. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to MDG1015 excipients, LDC agents, rasburicase, methylprednisolone or tocilizumab.
8. Untreated CNS metastases or active CNS metastases (progressing or requiring corticosteroids for symptoms control) and leptomeningeal disease
9. Unstable/active ulcer, varices, or digestive tract bleeding or recent digestive surgery that may have increased risk of bleeding
10. History of another primary malignancy that requires intervention beyond surveillance or that has not been in remission for at least 1 year. The following are exempt from the 1-year limit:

    1. non-melanoma skin cancer
    2. curatively treated localized prostate cancer
    3. carcinoma in situ (e.g. cervix, bladder, breast)
11. NYHA Class ≥ II, heart failure, unstable angina, a history of recent (≤ 6 months) arrythmias, myocardial infarction or sustained (> 30 seconds) ventricular tachyarrhythmias
12. Subjects who are dependent on dialysis
13. Subjects with a history of pulmonary embolism or deep vein thrombosis that cannot safely withhold anti-coagulant therapy from leukapheresis until 7 days after administration of MDG1015 as determined by the Investigator
14. Active autoimmune disease requiring systemic therapy except for adequately controlled Type 1 diabetes mellitus, autoimmune hypothyroidism or Grave's disease
15. Previous allogeneic hematopoietic stem cell transplant within the last 5 years or solid organ transplant

    Specific to GAC/GEJ Subjects:
16. Positive history of esophageal or gastric resection that the Investigator considers is at increased risk of bleeding or perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2042-08-01 (Estimated)

PRIMARY OUTCOMES:
DE Segment: Adverse Events and Dose Limiting Toxicities (Safety and Tolerability) | 28 days
  Incidence and severity of adverse events to establish RP2D measured by dose limiting toxicities (DLTs) up to 28 days post infusion
Exp Segment: Adverse Events (Safety) | 12 months
  Incidence of (S)AEs by type, grade and duration

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 months
  Proportion of Subjects having a confirmed complete response (CR) or partial response (PR) per RECIST v1.1
Correlation of blood levels and the onset and/or severity of IP-related toxicities | 12 months
  Correlation of certain blood levels in serum over time and any correlation between these levels and the onset and/or severity of IP-related toxicities
Clinical benefit rate (CBR) | 12 months
  Proportion of Subjects having a sustained confirmed stable disease (SD) or a confirmed PR or CR for any duration of time per RECIST v1.1
Overall survival (OS) | 15 years
  The interval between MDG1015 infusion and date of death by any cause
Assess feasibility of MDG1015 generation in study population | 2 years
  Number of MDG1015 products manufactured which comply with the pre-defined release specifications
Progression Free Survival (PFS) | 12 months
  The interval between MDG1015 infusion and date of disease progression or death per RECIST v1.1
Duration of response (DOR) | 12 months
  The interval between the first documented response following MDG1015 infusion until first documented disease progression or death
Best overall response (BOR) | 12 months
  The best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease (PD) the smallest measurements recorded since the treatment started)
Time to response (TTR) | 12 months
  The interval between MDG1015 infusion and first documented CR or PR per RECIST v1.1
Levels of MDG1015 in blood over time | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Dr. Zhen, MD, Principal Investigator — Fred Hutch Cancer Center
Locations (1):
- Fred Hutch Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided